CLINICAL TRIAL: NCT04714021
Title: CO2 vs Air Insufflation in Children Undergoing PEG (CO2pegA) - a Multicenter Double Blind RCT
Brief Title: CO2 vs Air Insufflation in Children Undergoing PEG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: European Society of Pediatric Gastroenterology, Hepatology and Nutrition (Other)
Responsible Party: Principal Investigator, Tadej Battelino, Professor of Pediatrics, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CO2pegA
Record Dates: First submitted 2021-01-12; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Gastrostomy
Keywords: children; endoscopy; CO2 insufflation
MeSH Terms: interventions — Air

STUDY DESIGN:
Intervention Model Description: * single step PEG technique group divided to co2 or air insufflation group during endoscopy
  * pull technique PEG group divided to co2 or air insufflation group during endoscopy
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single steep arm- CO2 insufflation (Experimental): PEG will be performed by single step technique and CO2 will be insufflated during the endoscopy
  Interventions: Other: CO2
- Single steep arm- air insufflation (Active Comparator): PEG will be performed by single step technique and air will be insufflated during the endoscopy
  Interventions: Other: air
- Pull technique arm- CO2 insufflation (Experimental): PEG will be performed by pull technique and CO2 will be insufflated during the endoscopy
  Interventions: Other: CO2
- Pull technique arm- air insufflation (Active Comparator): PEG will be performed by pull technique and air will be insufflated during the endoscopy
  Interventions: Other: air

INTERVENTIONS:
Other: CO2 — to insufflate CO2 into the stomach instead of air during the PEG
  Arms: Pull technique arm- CO2 insufflation; Single steep arm- CO2 insufflation
Other: air — to insufflate air into the stomach instead of CO2 during the PEG
  Arms: Pull technique arm- air insufflation; Single steep arm- air insufflation

SUMMARY:
Ap¬plications of CO2 insufflation for endoscopic procedures have been reported for the performance of routine colonoscopy, small bowel endoscopy, endoscopic retro¬grade cholangiopancreatography (ERCP) and endoscopic submucosal dissection in the upper and lower gastrointestinal tracts. These studies showed that CO2 insufflation reduces the post-procedural abdominal distension and pain without CO2 retention and adverse events. However, there has been no report on the safety and efficacy of CO2 insufflation in PEG procedures in adults or in children. In the present study, we would like to evaluate by randomized controlled trial: the safety of the CO2 insufflation during PEG and the inhibi¬tory effects of CO2 insufflation on bowel distension after PEG.

DETAILED DESCRIPTION:
Ap¬plications of CO2 insufflation for endoscopic procedures have been reported for the performance of routine colonoscopy, small bowel endoscopy, endoscopic retro¬grade cholangiopancreatography (ERCP) and endoscopic submucosal dissection in the upper and lower gastrointestinal tracts. These studies showed that CO2 insufflation reduces the post-procedural abdominal distension and pain without CO2 retention and adverse events. However, there has been no report on the safety and efficacy of CO2 insufflation in PEG procedures in adults or in children. In the present study, we would like to evaluate by randomized controlled trial: the safety of the CO2 insufflation during PEG and the inhibi¬tory effects of CO2 insufflation on bowel distension after PEG.

The primary objective is to determine the safety of the CO2 insufflation during PEG. The secondary objective of this study is to investigate the inhibitory effect of CO2 insufflation on bowel distension.

This is an investigator initiated multicentre, randomized, double blind study to evaluate the safety and adverse events profile of CO2 insufflation during PEG procedure. The study included a screening, pre-intervention (pre-PEG) and a post-intervention time (after-PEG), with total of 4 measurements of waist circumference, two measurements of i-stat.

Children aged 0-19 years, who were admitted for PEG procedure and who meet all inclusion and none of the exclusion criteria listed below. A total of 120 children after PEG insertion will be included and divided in two groups: one step group and standard pull group of children; two established groups will be randomized 1:1.

Inclusion criteria

* Male or female patients
* Age between 0 - 19 years
* Written informed consent Exclusion criteria
* Absolute contraindication for PEG procedure
* Patients with hypercapnia (pCO2 > 50 mmHg at first i-stat measurement)
* Language barriers which do not allow to give informed consent Patient data will be collected: age, gender, body mass index (BMI), underlining disease, duration of procedure, type of procedure, type of the scope, type of sedation or anaesthesia, complications.

Due to study protocol capillary blood will be withdrawn twice. To conclude there are actually no additional risks for included children due to the study protocol. Moreover, we will be able to diagnose early the important pneumoperitoneum, if it will occur and start to treat it with effective pain killers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients indicated for PEG procedure
* Age between 0 - 19 years
* Written informed consent

Exclusion Criteria:

* Absolute contraindication for PEG procedure
* Patients with hypercapnia (pCO2 > 50 mmHg at first i-stat measurement)
* Language barriers which do not allow to give informed consent

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2023-01-07 (Estimated); Study Completion 2023-01-07 (Estimated)

PRIMARY OUTCOMES:
To asses the change in pCO2 before and after the procedure | Time 0- (before the procedure) and at time 30 minutes (approximate end of procedure)
  Perform i-stat measurement (capillary pCO2 value in mmHg)

SECONDARY OUTCOMES:
To asses the change in waist circumference comparing CO2 and air insufflation | at four different time points: at time 0 (just before the procedure), 10 minutes later, 120 minutes later and 240 minutes later
  Perform waist measurements at the level of umbilicus with measuring tape in cm

CONTACTS AND LOCATIONS:
Overall Officials: Matjaz Homan, PhD, Principal Investigator — Children's Hospital in Ljubljana; Mike Thomson, PhD, Principal Investigator — Sheffield Children's Hospital
Locations (7):
- Paediatric Gastroenterology-Hepatology, Queen Fabiola Children's University Hospital, Brussels, Belgium
- Children's Hospital Zagreb, Zagreb, Croatia
- Policlinico Universitario Messina, Messina, Italy
- University Children's Hospital, Ljubljana, Slovenia
- University Children's Hospital Basel, Basel, Switzerland
- Al Jalila Children's Specialty Hospital, Dubai, United Arab Emirates
- Sheffield Children's Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
to use REDCap platform (gender, age, weight, BMI, type of procedure, type of anestesia, type of the endoscopy, time of PEG insertion, underlining diseases, complications, stat, waist circumference)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after finishing the study to main investigators (2 years) for 1 months
Access Criteria: principal investigators

REFERENCES:
- [Result] Gauderer MW, Ponsky JL, Izant RJ Jr. Gastrostomy without laparotomy: a percutaneous endoscopic technique. J Pediatr Surg. 1980 Dec;15(6):872-5. doi: 10.1016/s0022-3468(80)80296-x. PMID 6780678
- [Result] Thomson M, Rao P, Rawat D, Wenzl TG. Percutaneous endoscopic gastrostomy and gastro-oesophageal reflux in neurologically impaired children. World J Gastroenterol. 2011 Jan 14;17(2):191-6. doi: 10.3748/wjg.v17.i2.191. PMID 21245991
- [Result] Homan M, Mahkovic D, Orel R, Mamula P. Randomized, double-blind trial of CO2 versus air insufflation in children undergoing colonoscopy. Gastrointest Endosc. 2016 May;83(5):993-7. doi: 10.1016/j.gie.2015.08.073. Epub 2015 Sep 10. PMID 26363332
- [Result] Maple JT, Keswani RN, Hovis RM, Saddedin EZ, Jonnalagadda S, Azar RR, Hagen C, Thompson DM, Waldbaum L, Edmundowicz SA. Carbon dioxide insufflation during ERCP for reduction of postprocedure pain: a randomized, double-blind, controlled trial. Gastrointest Endosc. 2009 Aug;70(2):278-83. doi: 10.1016/j.gie.2008.12.050. Epub 2009 Jun 11. PMID 19523621